CLINICAL TRIAL: NCT01383252
Title: Comparison of Study Method Versus Conventional Method for Performing Unsedated Colonoscopy for Colorectal Cancer Screening and Surveillance
Brief Title: Unsedated Colonoscopy for Colorectal Cancer Screening and Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: VANCHCS-GI-005
Record Dates: First submitted 2011-06-21; First posted 2011-06-28 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Colon Polyp
Keywords: water method; air method; unsedated colonoscopy; adenoma detection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water method (Experimental): Water infusion in lieu of air insufflation for screening and surveillance colonoscopy
  Interventions: Procedure: Water infusion in lieu of air insufflation
- Air method (Active Comparator): Air insufflation for screening and surveillance colonoscopy
  Interventions: Procedure: Air method

INTERVENTIONS:
Procedure: Water infusion in lieu of air insufflation — Air pump is turned off, water is infused using a peristaltic pump to aid colonoscope insertion until the cecum is reached. Air pockets and dirty water are suctioned before clean water is infused (exchange) to facilitate scope insertion.
  Other Names: Water method; Screening colonoscopy
  Arms: Water method
Procedure: Air method — Conventional air method with minimal insufflation of air to aid scope insertion until the cecum is reached. Water in aliquots will be used for irrigation and cleansing.
  Other Names: Screening colonoscopy
  Arms: Air method

SUMMARY:
In a prospective, randomized, controlled study, two methods (water method vs. air method) of performing colonoscopy will be compared in patients undergoing unsedated colonoscopy for CRC screening. The investigators hypothesize that:

1. Study method increases overall cecal intubation with comparable assessment of current experience and patient willingness to repeat future colonoscopy compared with conventional colonoscopy
2. Study method improves bowel preparation and increases polyp pickup rate

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening for the high and the low risk healthy asymptomatic Veterans Affairs (VA) patients is being promoted. Compliance with this Directive will result in an increased number of VA patients undergoing colonoscopy.

The demand for colonoscopy far exceeds the capacity available to perform the procedure in the VA system. The conventional practice for colonoscopy at VA facilities across the country is to perform colonoscopy under conscious sedation with air insufflation. Efficiency is governed by the fact that sedated patients require time and space for recovery and these are major limiting factors in the current setting for the use of colonoscopy for CRC screening.

In a prospective, randomized, controlled trial (RCT), two methods of performing colonoscopy will be compared in patients undergoing unsedated colonoscopy for CRC screening. We compared the water infusion in lieu of air insufflation (water method) with the conventional air insufflation method. We hypothesize that the water method (Study method) increases overall cecal intubation with comparable assessment of current experience and patient willingness to repeat future colonoscopy compared with conventional colonoscopy. In addition, the water method improves bowel preparation and increases polyp pickup rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>50 years old)
* Male and female patients
* Scheduled and consented for screening or surveillance colonoscopy without medications
* Accept randomization to the study or the conventional method
* Agree to complete study questionnaires
* The adults will be normal healthy patients or patients with mild systemic disease, ASA 1 or ASA 2.

Exclusion Criteria:

* Patients who decline to participate
* Unable to give informed consent or complete the questionnaires due to language or other difficulties

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Success of colonoscopy | 24 months
  successful cecal intubation

SECONDARY OUTCOMES:
Polyp detection | 24 months
  Adenoma detection rate

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leung, MD, Principal Investigator — Sacramento VA Medical Center
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

REFERENCES:
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Background] Leung JW, Mann S, Leung FW. Options for screening colonoscopy without sedation: a pilot study in United States veterans. Aliment Pharmacol Ther. 2007 Aug 15;26(4):627-31. doi: 10.1111/j.1365-2036.2007.03404.x. PMID 17661766
- [Background] Leung FW, Mann SK, Salera R, Toomsen L, Cabrera H, Prather D, Gutierrez R, Leung JW. Options for screening colonoscopy without sedation: sequel to a pilot study in U.S. veterans. Gastrointest Endosc. 2008 Apr;67(4):712-7. doi: 10.1016/j.gie.2007.10.028. Epub 2008 Feb 14. PMID 18279868
- [Background] Leung JW, Salera R, Toomsen L, Mann S, Leung FW. Pilot feasibility study of the method of water infusion without air insufflation in sedated colonoscopy. Dig Dis Sci. 2009 Sep;54(9):1997-2001. doi: 10.1007/s10620-008-0576-4. Epub 2008 Dec 5. PMID 19058003